CLINICAL TRIAL: NCT00889096
Title: Effects of Propranolol on the Encoding and Retrieval of Emotional Material After Single Dose Administration in Healthy Young Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Prof. W. Siegmund, MD, Department of Clinical Pharmacology, Ernst-Moritz-Arndt-University Greifswald
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: BBEmoMem
Record Dates: First submitted 2009-04-27; First posted 2009-04-28 (Estimated); Last update posted 2015-06-29 (Estimated); Status verified 2009-04

CONDITIONS: Memory; Heart Rate; Skin Electric Conductance; Amylase; Propanolol
Keywords: memory; heart rate; skin conductance; α-amylase; propranolol; tolerability
MeSH Terms: interventions — Propranolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- study day 1 propanolol (Active Comparator): Oral administration of 80 mg propranolol (1 capsule containing two Obsidan® tablets: 2 x 40 mg propranolol) according to randomization list with 240 ml. Determination of blood pressure, heart rate over 4 hours and until return to the initial baseline values.
  Interventions: Drug: propranolol
- study day 1 placebo (Placebo Comparator): Oral administration of placebo (1 capsule containing two placebo tablets) according to randomization list with 240 ml. Determination of blood pressure, heart rate over 4 hours and until return to the initial baseline values.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: propranolol — Oral administration of 80 mg propranolol (1 gelatine capsules; content: 2 tablets of Obsidan® 40 mg Tablets) or placebo (1 gelatine capsules; content: 1 tablet placebo; microcrystalline cellulose, magnesium stearate, cellulose powder, lactose monohydrate) according to randomization list with 240 ml tap water.
  Arms: study day 1 propanolol
Drug: placebo — Oral administration of placebo (1 gelatine capsules; content: 1 tablet placebo; microcrystalline cellulose, magnesium stearate, cellulose powder, lactose monohydrate) according to randomization list with 240 ml tap water.
  Arms: study day 1 placebo

SUMMARY:
1. To evaluate the effects of a single oral (80 mg) dose of propranolol on the encoding of emotional pictures as assessed by peripheral physiological and electrocortical parameters in a healthy population.
2. To evaluate the effects of a single oral (80 mg) dose of propranolol on the retrieval of emotional pictures as assessed by electrocortical parameters in a healthy population.
3. To evaluate correlations between behavioral data and psychophysiological parameters.

DETAILED DESCRIPTION:
The main objective of the present study is to combine two lines of research investigating the interaction between emotional processing and memory performance and its modulation by beta-blockade. As has been suggested by aforementioned lesion, pharmacological and neuroimaging evidence, emotional stimuli are better remembered because they are better encoded.

In the ERP literature, there are a number of studies on emotion and memory, but few of them have investigated the modulatory effects of emotion on memory, focusing on either during stages of encoding (Palomba, Angrilli & Mini, 1997; Dolcos & Cabeza, 2002) or during memory retrieval of emotional and neutral material (Maratos & Rugg, 2001; Windmann & Kutas, 2001). It is assumed that emotionally arousing information gains privileged access to processing resources. This means that emotional arousing stimuli guide attention for more elaborated processing, leading to better memory formation.

Concerning pharmacological manipulations with ß-blockers, there is no existing ERP study that shows the effect of ß-blockade on encoding processes and memory retrieval of emotional pictures. Therefore, the current investigation was designed to test whether recall and recognition of emotional pictures can be reduced by administration of propranolol and whether this reduction in memory performance is correlated with changes in event-related potentials or peripheral physiological parameters (heart rate variability, heart rate, blood pressure and electrodermal response). As a surrogate for sympathetic activity and/or activation by noradrenaline, a salivary sample to measure activity of the alpha-amylase will be employed (van Stegeren, Rohleder, Everaerd & Wolf, 2006) In conclusion, we hypothesize (1) a memory advantage for emotionally arousing stimuli but not for emotionally neutral pictures. (2) ERP components associated with emotional effects and memory effects are pronounced for emotional stimuli. (3) Peripheral physiological parameters should also be pronounced for emotionally arousing stimuli. (4) Emotional processing and emotional memory will be impaired by the beta-blocker propranolol as indicated by behavioral data and psycho-physiological parameters.

ELIGIBILITY:
Inclusion Criteria:

* age: 18 - 35 years
* sex: male
* ethnic origin: Caucasian
* body weight: between 19 kg/m² and 27 kg/m² [calculated from weight (kg)/height2 (m2)]
* good health as evidenced by the results of the clinical examination, ECG, and laboratory check-up, which are judged by the clinical investigator not to differ in a clinical relevant way from the normal state
* written informed consent

Exclusion Criteria:

* obstructive lung disease (e.g. bronchial asthma)
* peripheral arterial circulatory disturbance
* any disturbance of impulse formation and conduction (e.g. sick sinus syndrome, SA or AV-blockade)
* bradycardia (< 50 beats/min)
* hypotension (systolic pressure < 90 mmHg)
* existing cardiac or hematological diseases and/or pathological findings, which might interfere with the drug's safety, tolerability, absorption and/or pharmacokinetics
* existing hepatic and renal diseases and/or pathological findings, which might interfere with the drug's safety, tolerability, absorption and/or pharmacokinetics
* existing gastrointestinal diseases and/or pathological findings, which might interfere with the drug's safety, tolerability, absorption and/or pharmacokinetics
* existing or further diseases of the CNS, especially epilepsy
* acute or chronic diseases which could affect absorption or metabolism
* history of any serious psychological disorder
* taking MAO inhibitors
* drug or alcohol dependence
* positive drug or alcohol screening
* smokers
* positive anti-HIV-test, HBs-Ag-test or anti-HCV-test
* volunteers who are on a diet which could affect the pharmacokinetics of the drug
* heavy tea or coffee drinkers (more than 1L per day)
* volunteers suspected or known not to follow instructions
* volunteers working night shifts
* volunteers who are in stressful periods or had undergone major life changes (e.g. death of a close family member in the past year)
* volunteers who are unable to understand the written and verbal instructions, in particular regarding the risks and inconveniences they will be exposed to as a result of their participation in the study
* participation in another clinical trial during this study
* less than 14 days after last acute disease
* any systemically available medication within 4 weeks prior to the intended first administration unless because of the terminal elimination half-life complete elimination from the body can be assumed for the drug and/or its primary metabolites
* repeated use of drugs during the last 4 weeks prior to the intended first administration, which can influence hepatic biotransformation (e.g. barbiturates, cimetidine, phenytoin, rifampicin)
* repeated use of drugs during the last 2 weeks prior to the intended first administration which affect absorption (e.g. laxatives, metoclopramide, loperamide, antacids, H2-receptor antagonists)
* known allergic reactions to the active ingredients used or to constituents of the pharmaceutical preparation
* subjects with severe allergies or multiple drug allergies

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Estimated)

PRIMARY OUTCOMES:
memory performance for pictures

SECONDARY OUTCOMES:
heart rate and heart rate variability
blood pressure
skin conductance and responses electrocortical activity
α-amylase activity in saliva
tolerability of propranolol

CONTACTS AND LOCATIONS:
Overall Officials: Werner Siegmund, Prof, Principal Investigator — Department of Clinical Pharmacology, Ernst-Moritz-Arndt-University Greifswald
Locations (1):
- Department of Clinical Pharmacology, Ernst-Moritz-Arndt-University Greifswald, Greifswald, Mecklenburg-Vorpommern, Germany